CLINICAL TRIAL: NCT03208218
Title: An Open-label, Randomized, Single Dose, Crossover Bioequivalent Study to Compare Pharmacokinetic Property of SYP-1512 Tab and Revlimid Cap, 25mg in Healthy Male Volunteers
Brief Title: Crossover Study to Compare Pharmacokinetic Property of SYP-1512 Tab and Revlimid Cap in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Collaborators: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIBE2016-02
Record Dates: First submitted 2017-06-25; First posted 2017-07-05 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Healthy, Male
Keywords: Evaluation of the pharmacokinetics equivalence; Healthy volunteers; Single dose over the period I and II(crossover); Healthy male volunteers
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYP-1512 (Experimental): Lenalidomide 25mg/tablet, PO, 1 tablet once daily for I&II D1(crossover)
  Interventions: Drug: SYP-1512
- Revlimid cap. (Active Comparator): Lenalidomide 25mg/capsule, po, 1 capsule once daily for period I&II D1(crossover)
  Interventions: Drug: Revlimid cap

INTERVENTIONS:
Drug: SYP-1512 — Lenalidomide 25mg/tablet, PO, 1 tablet once daily for I&II D1(crossover)
  Other Names: Lenalidomide 25mg
  Arms: SYP-1512
Drug: Revlimid cap — Lenalidomide 25mg/capsule, po, 1 capsule once daily for period I&II D1(crossover)
  Other Names: Lenalidomide 25mg
  Arms: Revlimid cap.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics equivalence and safety by comparing pharmacokinetics characteristics between the SYP-1512 Tab and Revlimid cap (25mg) when administered a single-dose to healthy male volunteers.

DETAILED DESCRIPTION:
Healthy volunteers are administrated single-dose over the period I and II (crossover) of SYP-1512 Tab and Revlimid cap (25mg) as of lenalidomide 25mg.

Every time before and after each medication, pharmacokinetic (PK) parameters and safety of SYP-1512 Tab and Revlimid cap (25mg) is performed using a blood sample and conducting some tests (vital signs, physical exam, ECG, laboratory test, etc.) respectively

ELIGIBILITY:
Inclusion Criteria:

1. Over 20aged in healthy males
2. Those who do not have congenital or chronic diseases or pathological symptoms based on screening.
3. The person who is determined to be the subject of the clinical laboratory test results such as hematology test, blood chemistry test, urine test, etc. set by the person in charge of the examination of the medical institution
4. BMI : 18-30
5. Those who have not donated blood within 2 weeks
6. Those without a history of gastrointestinal resection
7. Those who have no history of mental illness within the last 5 years
8. Agreement with written informed consent
9. Anyone who can follow and follow all scheduled admission and outpatient visits, dosing, clinical laboratory testing and subject compliance
10. If the partner is a woman of childbearing age who does not use the appropriate method of contraception (even if the man has undergone a vasectomy), while taking lenalidomide, during the interruption, for consenting to use condoms for 28 days after the last dose
11. In the vital sign measured in a sitting position, the systolic blood pressure ≤145 mmHg and ≥100 mmHg, the diastolic blood pressure ≤95 mmHg and ≥60 mmHg, the pulse rate> 40 and <100 times / minute
12. Electrocardiogram (ECG) of the 12-electrode, QTc ≤ 450 msec
13. Those who have agreed not to donate blood or plasma and semen for at least 28 days after taking this drug
14. If the contraceptive is withdrawn due to contraception or partner's pregnancy confirmation during testing. Those who agree to respond to follow-up within 6 months after pregnancy and after delivery

Exclusion Criteria:

1. Those taking drugs that significantly induce drug metabolizing enzymes within one month before screening (eg, barbiturate) or inhibit
2. Those taking medication that could affect the test within 10 days before screening
3. The person who is in charge of the examination of the medical institution (or the examining doctor who is delegated)
4. Those who have participated in the bioequivalence test or other clinical studies within 3 months prior to the administration of the test and administered the clinical trial drug
5. Persons with hypersensitivity to venous puncture
6. Screening Within the first 6 months, a person with a history of regular alcohol consumption as follows: 1 cup = 150 mL of wine or 360 mL of beer or 45 mL of distillate)
7. Patients with severe hepatic impairment
8. Patients who are hypersensitive to NSAIDs and other components of NSAID
9. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
10. Patients with renal impairment (Cockcroft-Gault-type creatinine clearance <50 mL / min)
11. Positive result of Serum test [RPR Ab (VDRL), HBsAg, HCV Ab, anti HIV (AIDS)]

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of the AUCt between SYP-1512 and Revlimid cap(25mg) | 0-24hours
  Bioequivalance of the AUCt between SYP-1512 and Revlimid cap(25mg)
Pharmacokinetics of the Cmax between SYP-1512 and Revlimid cap(25mg) | 0-24hours
  Bioequivalance of the Cmax between SYP-1512 and Revlimid cap(25mg)

SECONDARY OUTCOMES:
Pharmacokinetics of the AUCinf SYP-1512 and Revlimid cap (25mg) | 0-inf
  Bioequivalance of the AUCinf SYP-1512 and Revlimid cap (25mg)
Pharmacokinetics of the Tmax of SYP-1512 and Revlimid cap (25mg) | 0-24hours
  Bioequivalance of the Tmax of SYP-1512 and Revlimid cap (25mg)
Pharmacokinetics of the T1/2 of SYP-1512 and Revlimid cap (25mg) | 0-24hours
  Bioequivalance of the T1/2 of SYP-1512 and Revlimid cap (25mg)

IPD SHARING:
Plan to Share IPD: No